CLINICAL TRIAL: NCT00315991
Title: Parent-Child Co-Regulation of Pediatric Diabetes, Phase 2
Brief Title: Blood Glucose Awareness Training for Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None
Other Study IDs: 12202
Record Dates: First submitted 2006-04-18; First posted 2006-04-19 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: BG perception; hypoglycemic awareness; pediatric T1DM
MeSH Terms: conditions — Diabetes Mellitus, Type 1

ARMS (2):
- BGAT Intervention (Experimental): Blood Glucose Awareness Training for Parents
  Interventions: Behavioral: Blood Glucose Awareness Training for Parents
- Control (No Intervention): Enter PDA data and complete questionnaires only. No intervention received.

INTERVENTIONS:
Behavioral: Blood Glucose Awareness Training for Parents
  Arms: BGAT Intervention

SUMMARY:
The purpose of this study is to test a training program for parents of children with T1DM.

DETAILED DESCRIPTION:
Successful diabetes management relies on a process of self-regulation in which treatment behavior is guided by feedback about changing blood glucose (BG) levels and decision-making. The processes involved in self-regulation have been studied extensively in adults with Type 1 Diabetes Mellitus (T1DM), leading to the development of sophisticated research tools that have significantly advanced our understanding and ability to predict clinical outcome. Additionally, this research has led to the development of a highly effective, empirically based,pyschobehavioral intervention, Blood Glucose Awareness Training (BGAT) that improves self-regulation and clinical outcome in adults with T1DM. Unfortunately, the processes involved in the self-regulation of pediatric diabetes have received virtually no empirical attention. The purpose of this project is to correct the scientific neglect of the self-regulation in pediatric diabetes by adapting the conceptual and methodological tools used in adult studies to investigate the process of diabetes regulation by school-aged children (6-11 years) with T1DM and their parents and to develop and test an intervention to enhance the skills critical to this process.

ELIGIBILITY:
Inclusion Criteria:

* Parent/Guardian with primary responsibility for a child's diabetes management
* Child with T1DM between the ages 6 - 11 years.
* Duration of child's diabetes > 1 year
* Routine self-testing of child's BG > 2x day
* Intention to remain in the study's geographical region for the next 5 months
* Have a computer at home

Exclusion Criteria:

* Significant comorbidity in the child that could interfere with BG awareness or psychosocial status
* Medications taken by the child that interfere with symptom perception
* Psychiatric disorder in a parent or child
* Cognitive deficits/learning disabilities in the child that might preclude ability to complete the study protocol.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 77 (Actual)
Dates: Start 2006-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of blood glucose level estimation | 70 trials over a one month period
  Parents and children asked to report symptoms and give an estimated bg level. Later compared to actual bg levels to give an accuracy rating.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Gonder-Frederick, Ph.D., Principal Investigator — University of Virginia, Department of Psychiatric Medicine, Behavioral Medicine Research
Locations (2):
- United States (2):
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia